CLINICAL TRIAL: NCT00646776
Title: Study to Evaluate the Exposure of Rifabutin Administered in an Alternate Regimen in Combination With Atazanavir and Ritonavir Healthy Subjects
Brief Title: Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-360
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Antivirals/HIV
MeSH Terms: interventions — Rifabutin; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Rifabutin
- B (Active Comparator)
  Interventions: Drug: Rifabutin + Atazanavir + Ritonavir

INTERVENTIONS:
Drug: Rifabutin — Capsule, Oral, 150 mg, once daily, 11 Days
  Arms: A
Drug: Rifabutin + Atazanavir + Ritonavir — Capsules, Oral, 18 Days
  Rifabutin (150 mg, 2x/wk)
  Atazanavir (300 mg, once daily)
  Ritonavir (100 mg, once daily)
  Other Names: Reyataz
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the exposure of rifabutin (RIB) when administered with atazanavir and ritonavir (ATV/RTV)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 to 50 years old with a body mass index (BMI) of 18 to 32 kg/m²
* Prior to enrollment, subjects must have physical and laboratory test findings within the normal limits, and women of childbearing potential (WOCBP) must have a negative pregnancy test

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiogram (ECG) or clinical laboratory determinations
* Use of any prescription drugs or over-the-counter acid controllers within 4 weeks prior to study drug administration
* Use of any other drugs, including over-the-counter medications of herbal preparations within 1 week prior to study drug administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb Clinical Pharmacology Unit, Hamilton, New Jersey, United States

REFERENCES:
- [Derived] Zhang J, Zhu L, Stonier M, Coumbis J, Xu X, Wu Y, Arikan D, Farajallah A, Bertz R. Determination of rifabutin dosing regimen when administered in combination with ritonavir-boosted atazanavir. J Antimicrob Chemother. 2011 Sep;66(9):2075-82. doi: 10.1093/jac/dkr266. Epub 2011 Jun 28. PMID 21712242

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 85 enrolled participants, 52 participants did not receive the study drug (49 did not meet the study criteria and 3 were not needed as study was fully enrolled).
Groups:
- RIB 150 mg Once Daily (QD): Participants were administered an oral dose of rifabutin (RIB) 150 mg QD on Days 1 to 10. RIB was given in the morning within 5 minutes of completing a light meal. Participants were admitted to the clinical facility the evening prior to dosing (Day -1) and remained confined for the duration of the study.
- ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly: Participants were administered an oral dose of atazanavir/ritonavir (ATV/RTV) 300/100 mg QD on Days 1 to 17 and an oral dose of RIB 150 mg twice weekly on Days 1, 4, 8, 11 and 15. Study treatment was given in the morning within 5 minutes of completing a light meal. Participants were admitted to the clinical facility the evening prior to dosing (Day -1) and remained confined for the duration of the study.
Period: Overall Study
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Started | 15 (Treated on Day 1) | 18 (Treated on Day 1)
Completed | 14 | 5
Not Completed | 1 | 13
Not completed — Adverse Event | 1 | 9
Not completed — Investigator discretion | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly | Total
Number analyzed (Participants) | 15 | 18 | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (5) | 37 (9) | 36 (7)
Age, Customized [Number; unit: participants]
  <65 years | 15 | 18 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 10 | 14 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Other race comprises American Indian/Alaskan
  participants
    Caucasian | 9 | 5 | 14
    Black or African American | 3 | 12 | 15
    Asian | 2 | 0 | 2
    Other Race | 1 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is defined as the individual's body weight divided by the square of his or her height.
  kg/m^2 | 26.1 (3.2) | 26.6 (3.5) | 26.4 (3.3)
Height Continuous [Mean (Standard Deviation); unit: cm] | 173.7 (7.3) | 174.4 (10.0) | 174.1 (8.8)
Weight Continuous [Mean (Standard Deviation); unit: kg] | 79.1 (12.0) | 81.3 (14.9) | 80.3 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Average Area Under the Plasma Concentration-time Curve for 24 Hours (AUC24avg) for Rifabutin (RIB)
Description: AUC24avg is AUC(0-24 hour) following dosing on Day 10 for RIB 150mg once daily (QD); AUC24avg is the area under the plasma concentration-time curve in 1 dosing interval (AUC[TAU]) divided by the number of days over the sampling duration for ATV/RTV 300/100 mg QD+RIB 150 mg twice weekly, i.e. AUC(TAU)/7.
Time Frame: Pre-dose (0 hours [h]) on Days 6, 8, 10, and 11, and post-dose (1h,2h,3h,4h,6h,8h,12h) on Day 10 for RIB 150 mg QD; and pre-dose (0h) on Days 4, 8,11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of RIB as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: nanograms*hour /milliliters (ng*h/mL)
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 14 | 7
nanograms*hour /milliliters (ng*h/mL) | 1565 (528.49) [960.1 to 2948] | 2311 (507.99) [1738 to 3108]
Statistical Analysis 1: Comparison: RIB 150 mg Once Daily (QD) vs ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 1.477, 90% CI 2-sided [1.188 to 1.835] — Point estimates and 90% confidence intervals of treatment differences on the log scale were exponentiated to obtain estimates on the original scale

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of RIB
Description: Cmax was derived from plasma concentration versus time for RIB and was recorded directly from experimental observations for each treatment period.
Time Frame: Pre-dose (0h) on Days 6, 8, 10, and 11, and post-dose (1h,2h,3h,4h,6h,8h,12h) on Day 10 for RIB 150 mg QD; and pre-dose (0h) on Days 4, 8,11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of RIB as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 14 | 7
ng/mL | 159.0 (50.52) [109.3 to 262.0] | 395.6 (54.32) [322.0 to 469.3]
Statistical Analysis 1: Comparison: RIB 150 mg Once Daily (QD) vs ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 2.489, 90% CI 2-sided [2.025 to 3.060] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Minimum Plasma Concentration (Cmin) of RIB
Description: Cmin was derived from plasma concentration versus time for RIB.
Time Frame: as for outcome 2
Population: All treated participants who received all doses of RIB as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 14 | 7
ng/mL | 28.89 (14.08) [16.25 to 67.44] | 40.49 (11.27) [29.21 to 61.59]
Statistical Analysis 1: Comparison: RIB 150 mg Once Daily (QD) vs ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 1.402, 90% CI 2-sided [1.052 to 1.867] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax of ATV
Description: Cmax was derived from the plasma concentration versus time for ATV and was recorded directly from experimental observations for each treatment period.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of ATV as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly: Participants were randomized to receive Atazanavir/Ritonavir 300/100mg orally once daily on Days 1 to 17. Participants also received oral dose of Rifabutin 150 mg twice weekly on Days 1, 4, 8, 11 and 15. Participants were dosed in the morning within 5 minutes of completing a light meal. Participants were admitted to the clinical facility the evening prior to dosing (Day -1) and remained confined for the duration of the study.
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
ng/mL | 5633 (940.84) [4110 to 7130]
Statistical Analysis 1: Comparison: ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 0.947, 90% CI 2-sided [0.817 to 1.098]

5. Secondary Outcome: Cmin of ATV
Description: Cmin was derived from the plasma concentration versus time for ATV.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of ATV as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
ng/mL | 920.69 (497.07) [444.00 to 2190.00]
Statistical Analysis 1: Comparison: ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; p = 0.0963, ANOVA; Point Estimate = 0.7450, 90% CI 2-sided [0.5569 to 0.9967]

6. Secondary Outcome: AUC(TAU) for ATV
Description: AUC(TAU) was derived from the plasma concentration versus time for ATV, and was calculated by linear and log-linear trapezoidal summations using a mixed log-linear algorithm.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of ATV as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
ng*h/mL | 51795 (12680.65) [37082 to 83050]
Statistical Analysis 1: Comparison: ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 0.857, 90% CI 2-sided [0.723 to 1.015]

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of ATV
Description: Tmax was derived from the plasma concentration versus time for ATV and was recorded directly from experimental observations for each treatment period.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of ATV as specified per protocol, and were evaluable for analysis.
Measure: Median (Full Range); unit: Hour
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
Hour | 2.00 (0.88) [2.00 to 4.00]

8. Secondary Outcome: Terminal Elimination Half-life (T-half) of ATV
Description: T-half was obtained directly from the concentration-time data. T-half following doses administered for treatment ATV/RTV 300/100 mg QD+RIB 150 mg twice weekly.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of ATV as specified per protocol, and were evaluable for analysis.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
Hour | 11.89 (3.65) [7.58 to 18.98]

9. Secondary Outcome: Cmax of RTV
Description: Cmax was derived from the plasma concentration versus time for RTV and was recorded directly from experimental observations for each treatment period.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of RTV as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
ng/mL | 1466 (467.23) [830.0 to 2200]
Statistical Analysis 1: Comparison: ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 0.660, 90% CI 2-sided [0.538 to 0.809]

10. Secondary Outcome: Cmin of RTV
Description: Cmin was derived from the plasma concentration versus time for RTV.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of RTV as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
ng/mL | 40.54 (34.78) [20.80 to 130.0]
Statistical Analysis 1: Comparison: ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 0.651, 90% CI 2-sided [0.430 to 0.986]

11. Secondary Outcome: AUC(TAU) for RTV
Description: AUC(TAU) was derived from the plasma concentration versus time for RTV, and was calculated by linear and log-linear trapezoidal summations using a mixed log-linear algorithm.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of RTV as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
ng*h/mL | 8699 (3002.89) [5619 to 12999]
Statistical Analysis 1: Comparison: ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 0.696, 90% CI 2-sided [0.563 to 0.862]

12. Secondary Outcome: Tmax of RTV
Description: Tmax was derived from the plasma concentration versus time for RTV and was recorded directly from experimental observations for each treatment period.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of RTV as specified per protocol, and were evaluable for analysis.
Measure: Median (Full Range); unit: Hour
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
Hour | 4.00 (0.87) [3.00 to 6.00]

13. Secondary Outcome: T-half of RTV
Description: T-half was obtained directly from the concentration-time data.
Time Frame: Pre-dose (0h) on Days 4, 8, 11 to 18 and post-dose (1h,2h,3h,4h,6h,8h,12h) on Days 11 and 15 for ATV/RTV + RIB.
Population: All treated participants who received all doses of RTV as specified per protocol, and were evaluable for analysis.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 9
Hour | 4.45 (0.65) [3.52 to 5.66]

14. Secondary Outcome: Number of Participants Who Died, Experienced Other Serious Adverse Events (SAEs), Experienced Adverse Events (AEs) and Experienced Events Leading to Discontinuation.
Description: AEs were defined as new, untoward medical occurrences/worsening of pre-existing medical condition, whether drug-related or not. SAEs were defined as any AE that: resulted in death; was life threatening; resulted in a persistent or significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; was a cancer; or was an overdose. Discontinuation from the study was due either to an AE or was conducted at the investigator's discretion.
Time Frame: From Day 1 to 30 days after the last dose of study drug.
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants
  Deaths | 0 | 0
  Other SAEs | 0 | 2
  AEs | 5 | 13
  AE leading to discontinuation | 1 | 9
  Discontinuation due to investigator discretion | 0 | 4

15. Secondary Outcome: Number of Participants With Marked Abnormalities (MAs) in Hematology: Hemoglobin, Hematocrit, Platelet Count and Leukocytes
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Hemoglobin/hematocrit: <0.85 x pre-treatment (pre-Rx) value. Platelet count: <0.85 x lower limit of normal (LLN) (or, if pre-Rx value <LLN, then <0.85 x pre-Rx value) or >1.5 x upper limit of normal (ULN). Leukocytes: <0.9 x LLN or >1.2 x ULN (or, if pre-Rx value <LLN, then <0.85 x pre-Rx or >ULN. If pre-Rx value >ULN, then >1.15 x pre-Rx or <LLN).
Time Frame: Pre-dose on Day -1 and post-dose on Days 3, 7, 11, 14, 20 and 26 for RIB 150 mg QD; and pre-dose on Day -1 and post-dose on Days 3, 7, 11, 14 and 18 for ATV/RTV 300/100 mg QD + RIB 150 mg twice weekly.
Population: All treated participants. If a value had "not evaluable" in the dataset, then these participants were not counted (hemoglobin and hematocrit).
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants
  Hemoglobin | 0 | 1
  Hematocrit | 0 | 1
  Platelet count | 0 | 0
  Leukocytes | 1 | 7

16. Secondary Outcome: Number of Participants With MAs in Hematology: Neutrophils + Bands (Absolute), Lymphocytes (Absolute), Monocytes (Absolute), Basophils (Absolute) and Eosinophils (Absolute)
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Neutrophils+bands (absolute): <=1.50 x 10^3 cells/microliter (uL). Lymphocytes (absolute): <0.75 x 10^3 cells/uL or >7.50 x 10^3 cells/uL. Monocytes (absolute): >2.00 x 10^3 cells/uL. Basophils (absolute): >0.40 x 10^3 cells/uL. Eosinophils (absolute): >0.75 x 10^3 cells/uL.
Time Frame: as for outcome 15
Population: All treated participants. If a value had "not evaluable" in the dataset, then these participants were not counted(neutrophils + bands [absolute], monocytes [absolute], basophils [absolute] and eosinophils [absolute]).
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants
  Neutrophils+bands (absolute) | 1 | 10
  Lymphocytes (absolute) | 1 | 5
  Monocytes (absolute) | 0 | 0
  Basophils (absolute) | 0 | 0
  Eosinophils (absolute) | 0 | 0

17. Primary Outcome: AUC24avg for 25-O-Desacetyl-RIB
Description: AUC24avg is AUC(0-24 hour) following dosing on Day 10 for RIB 150 mg QD; AUC24avg is the area under the plasma concentration-time curve in 1 dosing interval (AUC[TAU]) divided by the number of days over the sampling duration for ATV/RTV 300/100 mg QD+RIB 150 mg twice weekly, i.e. AUC(TAU)/7
Time Frame: as for outcome 2
Population: All treated participants who received all doses of RIB as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 14 | 7
ng*h/mL | 117.7 (53.48) [46.0 to 240.7] | 1283 (260.71) [842.0 to 1634]
Statistical Analysis 1: Comparison: RIB 150 mg Once Daily (QD) vs ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 10.902, 90% CI 2-sided [8.135 to 14.610]

18. Primary Outcome: Cmax of 25-O-Desacetylrifabutin (25-O-Desacetyl-RIB)
Description: Cmax was derived from the plasma concentration versus time for 25-O-Desacetyl-RIB (a metabolite of RIB) and was recorded directly from experimental observations for each treatment period.
Time Frame: as for outcome 2
Population: All treated participants who received all doses of RIB as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 14 | 7
ng/mL | 13.44 (4.50) [7.14 to 22.10] | 104.36 (21.31) [64.21 to 128.3]
Statistical Analysis 1: Comparison: RIB 150 mg Once Daily (QD) vs ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANCOVA; Point Estimate = 7.766, 90% CI 2-sided [6.133 to 9.833]

19. Primary Outcome: Cmin of 25-O-Desacetyl-RIB
Description: Cmin was derived from plasma concentration versus time for 25-O-Desacetyl-RIB.
Time Frame: as for outcome 2
Population: All treated participants who received all doses of RIB as specified per protocol, and were evaluable for analysis.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 14 | 7
ng/mL | 2.79 (1.40) [2.03 to 5.42] | 31.97 (10.60) [22.13 to 53.44]
Statistical Analysis 1: Comparison: RIB 150 mg Once Daily (QD) vs ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 11.451, 90% CI 2-sided [8.147 to 16.095]

20. Primary Outcome: Total Area Under the Plasma Concentration-time Curve (AUCtot)
Description: AUCtot represents the total free RIB plus 25-O-Desacetyl-RIB output. It is calculated as: AUCtot (micromolar[µM]*h) = AUC24avg(RIB)(ng*h/mL)/847.016 (g/mole) + AUC24avg(25-O-Desacetyl-RIB)(ng*h/mL)/804.979(g/mole). The 300 mg RIB arm represents an extrapolation from the 150 mg RIB group.
Time Frame: as for outcome 2
Population: All treated participants who received all doses of RIB as specified per protocol, and were evaluable for analysis. The RIB 300 mg arm represents an extrapolation of the RIB 150 mg arm and as such, does not have a value for "Number of Participants Analyzed". AUCtot for RIB 300 mg QD was calculated as 2 × AUCtot for RIB 150 mg QD.
Measure: Geometric Mean (Full Range); unit: µM*h
Groups:
- ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly: Participants were administered an oral dose of atazanavir/ritonavir (ATV/RTV) 300/100 mg QAD on Days 1 to 17 and an oral dose of RIB 150 mg twice weekly on Days 1, 4, 8, 11 and 15. Study treatment was given in the morning within 5 minutes of completing a light meal. Participants were admitted to the clinical facility the evening prior to dosing (Day -1) and remained confined for the duration of the study.
- RIB 300 mg QD: AUCtot for RIB 300 mg QD was calculated as 2 × AUCtot for RIB 150 mg QD.
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly | RIB 300 mg QD
Number analyzed (Participants) | 14 | 7 | 0
µM*h | 2.00 (0.68) [1.19 to 3.77] | 4.38 (0.57) [3.52 to 5.35] |
Statistical Analysis 1: Comparison: RIB 150 mg Once Daily (QD) vs ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly; Test type: Superiority or Other; ANOVA; Point Estimate = 2.190, 90% CI 2-sided [1.783 to 2.691] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Number of Participants With MAs in Serum Chemistry: Alkaline Phosphatase (ALP),Aspartate Aminotransferase (AST),Alanine Aminotransferase (ALT),Bilirubin (Total),Bilirubin (Direct),Blood Urea Nitrogen (BUN),Creatinine,Sodium (Serum),Potassium (Serum)
Description: MAs=laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria. ALP, AST, ALT:>1.25xULN (if pre-Rx >ULN, then >1.25xpre-Rx). Bilirubin (total), bilirubin (direct), BUN:>1.1xULN (if pre-Rx >ULN, then >1.25xpre-Rx). Creatinine:>1.33xpre-Rx. Sodium (serum):<0.95xLLN or >1.05xULN (if pre-Rx <LLN, then <0.95xpre-Rx or >ULN. If pre-Rx >ULN, then >1.05xpre-Rx or <LLN). Potassium (serum):<0.9xLLN or >1.1xULN (if pre-Rx <LLN, then <0.9xpre-Rx or >ULN. If pre-Rx >ULN, then >1.1xpre-Rx or <LLN).
Time Frame: as for outcome 15
Population: All treated participants. If a value had "not evaluable" in the dataset, then these participants were not counted (ALP, AST, ALT, bilirubin [total], bilirubin [direct], BUN and creatinine).
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants
  ALP | 0 | 0
  AST | 0 | 0
  ALT | 0 | 0
  Bilirubin (total) | 0 | 17
  Bilirubin (direct) | 0 | 16
  BUN | 0 | 0
  Creatinine | 0 | 1
  Sodium (serum) | 0 | 0
  Potassium (serum) | 0 | 0

22. Secondary Outcome: Number of Participants With MAs in Serum Chemistry: Chloride (Serum), Calcium (Total), Protein (Total), Bicarbonate, Phosphorous (Inorganic)
Description: MAs=laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria. Chloride (serum), calcium (total), protein (total):<0.9xLLN or >1.1xULN (if pre-Rx <LLN, then <0.9xpre-Rx or >ULN. If pre-Rx >ULN, then >1.1xpre-Rx or <LLN). Bicarbonate:<0.8xLLN or >1.2xULN (if pre-Rx value <LLN, then <0.8xpre-Rx value or >ULN. If pre-Rx >ULN, then >1.2xpre-Rx value or <ULN). Phosphorous (inorganic):<0.85xLLN or >1.25xULN (if pre-Rx <ULN, then <0.85xpre-Rx or <ULN. If pre-Rx >ULN, then >1.25x re-Rx or <LLN).
Time Frame: as for outcome 15
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants
  Chloride (serum) | 0 | 0
  Calcium (total) | 0 | 0
  Protein (total) | 0 | 0
  Bicarbonate | 0 | 0
  Phosphorous (inorganic) | 0 | 0

23. Secondary Outcome: Number of Participants With MAs in Serum Chemistry: Glucose (Fasting Serum), Albumin, Creatine Kinase, Uric Acid, Lactate Dehydrogenase (LDH)
Description: MAs=laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria. Glucose (fasting serum): <0.8 x LLN or >1.5 ULN (if pre-Rx <LLN, then <0.8 x pre-Rx or >ULN. If pre-Rx >ULN, then >2.0 x pre-Rx or <LLN. Albumin: <0.9 x LLN (if pre-Rx <LLN, then <0.9 x pre-Rx). Creatine kinase: >1.5 x ULN (if pre-Rx >ULN, then >1.5 x pre-Rx). Uric acid: >1.2 x ULN (if pre-Rx >ULN, then >1.25 x pre-Rx). LDH: >1.25 x ULN (if pre-Rx >ULN, then >1.5 x pre-Rx).
Time Frame: as for outcome 15
Population: All treated participants. If a value had "not evaluable" in the dataset, then these participants were not counted(albumin, creatine kinase, uric acid and LDH).
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants
  Glucose (Fasting Serum) | 0 | 0
  Albumin | 0 | 0
  Creatine Kinase | 0 | 0
  Uric Acid | 0 | 0
  LDH | 0 | 0

24. Secondary Outcome: Number of Participants With MAs in Urinalysis
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following definitions specify the criteria for MAs. Protein, glucose and blood: >=2+ (or, if pre-treatment value >=1+, then >= 2 x pre-treatment value).
Time Frame: Pre-dose on Day -1, Day 7 and discharge.
Population: All participants who received the study drug on Day 1 were included in the analysis. If a value had "not evaluable" in the dataset, then these participants were not counted (for all parameters: protein, glucose and blood).
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants
  Protein | 0 | 1
  Glucose | 0 | 0
  Blood | 0 | 1

25. Secondary Outcome: Number of Participants With Identified Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities were defined as findings that are clinically meaningful as judged by the investigator. A 12-lead ECG was recorded at least 5 minutes after the participant had been lying down and all ECG recordings were evaluated by the investigator. Abnormalities, if present at any study time point, were listed.
Time Frame: Pre-dose on Day -1 and study discharge.
Population: All participants who received the study drug on Day 1 were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants | 0 | 3

26. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs or Physical Examination Findings
Description: Vital signs assessments and physical examination were conducted throughout the study. Vital signs assessments included body temperature, respiratory rate, blood pressure (systolic and diastolic), and heart rate. Physical examination included a neurological examination (if ocular signs or symptoms occurred, a reflex to slit lamp exam was performed by an ophthalmologist). The investigator used his/her clinical judgment to decide whether or not abnormalities in vital signs or physical examination were clinically meaningful.
Time Frame: Vital signs:screening, prior to dosing on Day 1, Day 7, study discharge. Physical examination:screening, Day -1, Day 7, study discharge
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | RIB 150 mg Once Daily (QD) | ATV/RTV 300/100 mg QD+RIB 150 mg Twice Weekly
Number analyzed (Participants) | 15 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | ATV/RTV 300/100mg+RIB 150mg | RIB 150mg
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/15
Other Adverse Events (participants affected / at risk) | 13/18 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV 300/100mg+RIB 150mg (N=18) | RIB 150mg (N=15)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV 300/100mg+RIB 150mg (N=18) | RIB 150mg (N=15)
PALPITATIONS (Cardiac disorders) | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0
EYE PAIN (Eye disorders) | 1 | 0
EYE PRURITUS (Eye disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 0
DRY MOUTH (Gastrointestinal disorders) | 1 | 0
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 1
LIP SWELLING (Gastrointestinal disorders) | 1 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 0
CHILLS (General disorders) | 2 | 1
FATIGUE (General disorders) | 1 | 0
FEELING COLD (General disorders) | 1 | 0
PAIN (General disorders) | 3 | 1
PYREXIA (General disorders) | 6 | 1
JAUNDICE (Hepatobiliary disorders) | 3 | 0
CELLULITIS (Infections and infestations) | 1 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 5 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 2
DIZZINESS (Nervous system disorders) | 3 | 0
HEADACHE (Nervous system disorders) | 3 | 2
HYPOAESTHESIA (Nervous system disorders) | 1 | 0
SLEEP DISORDER (Psychiatric disorders) | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 2 | 0
CHOKING SENSATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 2
FLUSHING (Vascular disorders) | 1 | 0
HOT FLUSH (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.